CLINICAL TRIAL: NCT04169776
Title: Effect of Daily Transcutaneous Auricular Vagus Nerve (taVNS) Stimulation on Proteinuria in Pediatric Patients With Idiopathic Nephrotic Syndrome
Brief Title: Effect of Daily Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) on Proteinuria in Pediatric Patients With Idiopathic Nephrotic Syndrome
Acronym: taVNS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: 19-0861
Record Dates: First submitted 2019-11-15; First posted 2019-11-20 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Idiopathic Nephrotic Syndrome; Frequently Relapsing Nephrotic Syndrome
MeSH Terms: conditions — Nephrosis, Lipoid; Nephrotic Syndrome

STUDY DESIGN:
Intervention Model Description: This study is a prospective cohort pilot study not formally classified as a specific trial phase. The study will involve two Arms, with 15 participants in each Arm of the study. Arm 1 will recruit patients with steroid-sensitive frequently-relapsing idiopathic nephrotic syndrome. Arm 2 will recruit patients with steroid-resistant idiopathic nephrotic syndrome. All participants in both Arms of the study will perform daily transcutaneous auricular vagus nerve stimulation (taVNS) therapy for 5 minutes each day. The study period will be 6 months. The participants will be monitored for labwork and clinical evidence of nephrotic syndrome relapse, comparing the number of relapses and level or proteinuria in the 6 months before starting taVNS therapy to number of relapses and level of proteinuria in the 6 month study period.
Masking Description: This study design was chosen as it is the most realistic and practical design for this pilot study. There is no blinding or masking in this pilot study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Steroid Sensitive Frequently-Relapsing Nephrotic Syndrome (Experimental): Individuals in this arm of the study will have to have a diagnosis of steroid sensitive frequently relapsing idiopathic nephrotic syndrome. They will receive transcutaneous auricular VNS (taVNS) performed for 5minutes every day for 6 months. The settings of the taVNS device will be individualized for each patient. Data will be collected on the the number of nephrotic syndrome relapses, the time between relapses, the time to remission once relapsed, and the level of proteinuria before and while using taVNS therapy.
  Interventions: Device: Transcutaneous Auricular Vagus Nerve (taVNS) stimulation
- Steroid Resistant Idiopathic Nephrotic Syndrome (Experimental): Individuals in this arm of the study will have to have a diagnosis of steroid resistant idiopathic nephrotic syndrome. They will receive transcutaneous auricular VNS (taVNS) performed for 5minutes every day for 6 months. The settings of the taVNS device will be individualized for each patient. Data will be collected on the the number of nephrotic syndrome relapses, the time between relapses, the time to remission once relapsed, and level of proteinuria before and while using taVNS therapy.
  Interventions: Device: Transcutaneous Auricular Vagus Nerve (taVNS) stimulation

INTERVENTIONS:
Device: Transcutaneous Auricular Vagus Nerve (taVNS) stimulation — Participants in this study will perform home transcutaneous auricular vagus nerve stimulation (taVNS) for 5 minutes a day for a 6-month period. The device that will be used is the commercially available Roscoe Medical TENS 7000 vagus nerve stimulator. The device will be attached to the Cymba Concha of the ear via an electrode ear clip. The intensity of the stimulation will be slowly increased and adjusted to individual tolerability for each treatment. TaVNS will be performed for 5 minutes daily for a period of 6 months.

SUMMARY:
This study evaluates the impact of transcutaneous auricular Vagus Nerve stimulation (taVNS) therapy on the incidence of nephrotic syndrome relapses in children with idiopathic nephrotic syndrome. Participants will perform taVNS 5 minutes a day for 6 months total, monitoring for signs of nephrotic syndrome relapse with both labwork and clinical symptoms.

DETAILED DESCRIPTION:
Idiopathic nephrotic syndrome is defined as the development of proteinuria, edema, hypoalbuminemia, and hyperlipidemia often presenting in the pediatric population. The underlying pathogenesis of idiopathic nephrotic syndrome is poorly understood but likely involves dysregulation of the immune system, and the majority of patients respond to steroid therapy and other immunosuppressive therapy. Unfortunately, relapses are common, with at least one relapse occurring in up to 90% of patients. Frequently-relapsing patients may be exposed large amounts of steroids and other immunosuppressants with a multitude of adverse effects, while others may not even respond to these treatments. Therefore, novel therapies are being studied.

Vagus nerve stimulation is a novel therapy with the potential to treat inflammatory conditions via inhibition of cytokine release by the cholinergic anti-inflammatory pathway. The purpose of the proposed study is to investigate the use of vagus nerve stimulation in the prevention of nephrotic syndrome relapses and treatment of proteinuria in pediatric patients with idiopathic nephrotic syndrome.

Patients will be enrolled if they have frequently-relapsing idiopathic nephrotic syndrome or proteinuria which does not respond to steroid therapy. These patients will perform daily transcutaneous auricular Vagus Nerve stimulation (taVNS) therapy 5 minutes a day for a 6 month period and will be monitored for urine/bloodwork or clinical signs of nephrotic syndrome relapse.

ELIGIBILITY:
Inclusion Criteria (Arm 1):

1. Subjects age 2-21 years of age
2. eGFR > 60 ml/min/1.73 m2
3. Diagnosis of idiopathic minimal change disease (clinical diagnosis or per biopsy)
4. Prior history of remission of nephrotic syndrome within 4 weeks of initiation of steroid therapy (steroid sensitive nephrotic syndrome)
5. 2 or more episodes of nephrotic syndrome relapses in a 6-month period or four or more episodes of nephrotic syndrome relapses in a 12-month period (relapse defined as 2+ proteinuria on first morning urine sample for three consecutive days or development of edema)
6. In remission (no proteinuria - normal urine protein to creatinine ratio < 0.2) at the time of enrollment

Inclusion Criteria (Arm 2):

1. Subjects age 2-21 years of age
2. eGFR > 60 ml/min/1.73 m2
3. Diagnosis idiopathic nephrotic syndrome (clinical diagnosis or per biopsy)
4. Diagnosis of steroid-resistant nephrotic syndrome (symptoms or proteinuria not improved after 4 to 8 weeks of steroid therapy)
5. Persistent proteinuria (first-morning urine protein to creatinine ratio > 0.2)
6. At least 7 days since last dose of steroids

Exclusion Criteria (Arm 1):

1. Subjects with nephrotic syndrome etiology other than idiopathic minimal change disease either biopsy-proven or by genetic testing
2. Nephrotic syndrome due to secondary causes such as SLE, vasculitis, hepatitis, post-infectious etiology, medication-induced, etc.
3. Subjects that did not achieve remission of nephrotic syndrome within 4 weeks of initiation of steroid therapy (steroid-resistant nephrotic syndrome)
4. Subjects with urine protein to creatinine ratio of > 0.2 (not in remission)
5. Subjects currently receiving any standing immunosuppressive therapy (mycophenolate mofetil, tacrolimus, rituximab - note: 1) previous exposure to these therapies does not exclude participation; 2) subjects with previous exposure to rituximab are eligible if B cells are replete)
6. Subjects with a history of cardiac issues, including bradycardia, arrhythmias or structural abnormalities of the heart
7. Subjects with implantable electronic devices such as pacemakers, defibrillators, hearing aids, cochlear implants or deep brain stimulators
8. Subjects with any other known inflammatory condition (IBD, SLE, etc.)

Exclusion Criteria (Arm 2):

1. Nephrotic syndrome due to secondary causes such as SLE, vasculitis, hepatitis, post-infectious etiology, medication-induced, etc.
2. Subjects with a history of cardiac issues, including bradycardia, arrhythmias or structural abnormalities of the heart
3. Subjects with implantable electronic devices such as pacemakers, defibrillators, hearing aids, cochlear implants or deep brain stimulators
4. Subjects with any other known inflammatory condition (IBD, SLE, etc.)

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of taVNS (Arms 1 and 2) | 6 months
  The endpoint of heart rate monitoring as a measure of safety of taVNS in this population was selected as this is the most concerning adverse effect of taVNS therapy. If there is no heart rate-related events during this study, it would further justify safe use of taVNS in the pediatric population.
  Tolerability is an important measure in this study but is mostly a subjective measure. Therefore, patients who withdraw due to intolerability or report side effects which are deemed intolerable will aid in determining the feasibility of taVNS use in this population.

SECONDARY OUTCOMES:
Impact of taVNS on cytokine levels (Arms 1 and 2) | 6 months
  TaVNS has been shown in literature to have an anti-inflammatory effect when stimulating the vagus nerve. Several studies have found that cytokine levels are increased in nephrotic syndrome relapses as compared to levels when in remission. This endpoint provides a measure of the efficacy and compliance of taVNS use while also providing a marker for the effect of taVNS on the patient. Finally, if taVNS is shown to reduce the number of relapses while also suppressing cytokine levels, it may suggest a cytokine-associated etiology of idiopathic nephrotic syndrome.
Impact of taVNS on number of nephrotic syndrome relapses, time to nephrotic syndrome relapses, and time to remission (Arm 1) | 6 months
  This outcome was chosen as an important measure of the efficacy of taVNS on patients with idiopathic nephrotic syndrome. A reduction in the number of relapses suggests that taVNS is a potential therapy for idiopathic nephrotic syndrome.
Impact of taVNS on level of proteinuria (Arm 2) | 6 months
  The marker of disease progression and worsening outcomes is the level of proteinuria in patients with steroid-resistant idiopathic nephrotic syndrome. Measurement of the urine protein to creatinine level on a first morning sample is the most feasible and accurate measure of proteinuria in this patient population.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Sethna, MD, Principal Investigator — Northwell Health
Locations (1):
- Northwell, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared if requested.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: 12/1/22 - ongoing
Access Criteria: Contact PI for data.

REFERENCES:
- [Derived] Merchant K, Zanos S, Datta-Chaudhuri T, Deutschman CS, Sethna CB. Transcutaneous auricular vagus nerve stimulation (taVNS) for the treatment of pediatric nephrotic syndrome: a pilot study. Bioelectron Med. 2022 Jan 26;8(1):1. doi: 10.1186/s42234-021-00084-6. PMID 35078538